CLINICAL TRIAL: NCT02799966
Title: Recovery of Upper Limb Function in Persons With Spinal Cord Injury: Lead-In Study
Acronym: MyndMove
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Collaborator, MyndTec, withdrew from the study due to lack of resources
Sponsor: University of British Columbia (Other)
Collaborators: Rick Hansen Institute (Other); MyndTec Inc. (Industry)
Responsible Party: Principal Investigator, Andrea Townson, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-00552
Record Dates: First submitted 2016-05-25; First posted 2016-06-15 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Traumatic Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Treatment Group (Other): Initiate treatment with MyndMove device on or after 10 days to 6 months (182 days) post spinal cord injury
  Interventions: Device: Myndmove
- Late Treatment Group (Other): Initiate treatment with MyndMove device on or after 6 months plus one day (183 days+) post spinal cord injury
  Interventions: Device: Myndmove

INTERVENTIONS:
Device: Myndmove — 20 sessions of 1 hour treatments with the MyndMove device (functional electrical stimulation) to the muscles of the upper limb(s), conducted 3 to 5 times per week, over 4 to 7 weeks.

SUMMARY:
Many individuals with cervical spinal cord injury (SCI) have difficulty using their hands and arms. MyndMove is a non-invasive medical device that uses short, low energy electrical pulses with surface electrodes to cause muscle contractions to produce a full range of reaching and grasping movements, which the patient is unable to perform by him/herself.

By using MyndMove therapy to help the individual move their arms and hands as he/she attempts to carry out typical reaching and grasping movements, the individual improves their ability to perform these tasks voluntarily.

The purpose of this study is to study the effectiveness of MyndMove therapy in improving the ability of individuals to move their arms and hands.

DETAILED DESCRIPTION:
There is no control group for this study. Participants from both treatment groups:

* Early treatment group = 10 days to 6 months post tSCI and
* Late treatment group = 6 months plus one day post tSCI

will receive one session (60 minutes) of MyndMove therapy, 3 to 5 times per week (only once per day), to gain 20 hours of intervention (total treatment duration will be 4 to 7 weeks).

Each 1 hour session includes therapy for single-arm or bilateral (left and right upper extremities) as clinically indicated for each study participant. Over the course of 20 one hour sessions, participants will progress through the various movement sequences aimed at regaining natural, unassisted voluntary movement in the affected limb(s). The MyndMove therapy will be in addition to the conventional upper limb rehabilitation therapy the participant will be prescribed to undertake at their local institution.

From previous experience, the first signs of function recovery may be expected to emerge two to four weeks after the onset of the MyndMove therapy program. As soon as the participant shows signs of recovery of either the voluntary extension or flexion in a stimulated muscle group, s/he will be encouraged to make an effort to voluntarily produce the movement that was previously facilitated by FES. As the participant demonstrates improved strength and range of motion, the FES for that muscle group will be phased out, and moved to another muscle group that is still paralyzed and needs to be "reactivated". The order in which muscle groups will be sequentially "reactivated" will be patient dependent.

Muscle reactivation milestones will be monitored and recorded during MyndMove therapy. The number of MyndMove treatments required to reach each milestone will be recorded. In addition, the overall time required to reach each milestone will be recorded.

Total duration of study participation, including a follow-up assessment, will be approximately 4 to 5 months.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic incomplete (AIS B-D) C4-C7 SCI
2. Early treatment group = 10 days to 6 months (182 days) post tSCI (note it is expected that most ppts will be recruited from this group, while at GF Strong)
3. Late treatment group = initiate treatment on or after 6 months plus one day (183 days+) post tSCI
4. SCIM self-care sub-score ≤ 10
5. Able to understand and follow instructions
6. Able to be in a seated position for a least one hour of upper limb therapy
7. Able to attend the study treatment sessions
8. Able to provide informed consent
9. Men and women of the age of majority in their province or state

Exclusion Criteria:

1. Previous history of any other neurological disorder or conditions that may affect motor response
2. Upper extremity injury or condition prior to SCI that limits the function of the hand or arm
3. Malignant skin lesion on the affected upper extremity
4. History of seizure disorder not effectively managed by seizure medications
5. An existing electrical stimulation devices (e.g. ICD, Pacemaker, Spinal Stimulation)
6. Rash or open wound at any potential electrode site
7. Denervation of muscles that are targeted by MyndMove
8. Poorly controlled autonomic dysreflexia (as determined by the local site physician)
9. In the judgment of the local site physician, participant has medical complications that may interfere with the execution of the study
10. Botulinum toxin injection into affected upper extremity within 3 months prior to the study start. No botulinum toxin injections during the study treatment and follow up period.
11. Currently enrolled in another upper limb study
12. Enrolled, in the past six months, in a clinical study involving drugs or biologics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Change in participant's ability to do regular tasks of daily living as measured by the Spinal Cord Independence Measure (SCIM) questionnaire | Change from baseline to 4/7 weeks
  This is a disability scale that has been specifically developed to evaluate the functional outcomes of patients with traumatic and non-traumatic SCI. The SCIM assesses function in three core areas: 1) Self-care, which includes feeding, bathing, dressing and grooming; 2) Respiration and sphincter management; and lastly 3) Mobility.
Change in participant's upper limb and hand impairment and function using GRASSP (Graded Refined Assessment of Strength Sensibility Test). | Change from baseline to 4/7 weeks
  This is a multi-modality test designed to assess the integration of sensorimotor hand and upper limb impairment and function. This test combines the features of several other tests that have been used to assess hand and upper limb function in the peripheral hand population.
Change in participant's reaching and grasping function with the Toronto Rehab Institute Hand Function Test (TRI-HFT). | Change from baseline to 4/7 weeks
  A test developed to evaluate improvements in the gross motor function of the unilateral grasp due to FES for reaching and grasping treatment. Hand functions that will be tested with the TRI-HFT are: lateral or pulp pinch, and palmar grasps.
Change in participant's grasp, grip, pinch and gross movement of the arm and upper limb using the Action Research Arm Test (ARAT). | Change from baseline to 4/7 weeks
  A test developed to assess the upper limb function in stroke and SCI patients. It consists of four sub-tests: grasp, grip, pinch and gross movement.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Townson, MD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - GF Strong Rehab Centre, Vancouver, British Columbia
  - Stan Cassidy Centre, Fredericton, New Brunswick
  - Toronto Rehabilitation Institute, Toronto, Ontario